CLINICAL TRIAL: NCT06795802
Title: Effect of Evaluative Conditioning on the Intensity of Physical Activity of Patients in a Cardiac Rehabilitation Program
Brief Title: Effect of Evaluative Conditioning on Intensity of Physical Activity of Patients Doing Cardiac Rehabilitation
Acronym: Cardio'Activ
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2023/AP-01
Record Dates: First submitted 2025-01-20; First posted 2025-01-28 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular Rehabilitation; Motivation; Physical Activity
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diet group: Patients in this group will receive Evaluative Conditioning favorable to diet. The evaluative conditioning procedure is a learning technique performed on a monitor. It consists of being exposed to the repeated association of an object (conditioned stimulus; in this case, fruit and vegetables) to stimuli with a positive or negative valence (unconditioned stimulus). The total duration of the Evaluative Conditioning is approximately 15 minutes.
  Interventions: Behavioral: Evaluative conditioning
- Physical Activity group: Patients in this group will receive Evaluative Conditioning favorable to Physical Activity. Patients in this group will receive Evaluative Conditioning favorable to diet. The evaluative conditioning procedure is a learning technique performed on a monitor. It consists of being exposed to the repeated association of an object (conditioned stimulus; in this case, Physical Activity) to stimuli with a positive or negative valence (unconditioned stimulus). The total duration of the Evaluative Conditioning is approximately 15 minutes.
  Interventions: Behavioral: Evaluative conditioning

INTERVENTIONS:
Behavioral: Evaluative conditioning — The evaluative conditioning procedure is a learning technique performed on a monitor. It consists of being exposed to the repeated association of an object (conditioned stimulus, in our case, Physical Activity or fruit and vegetables) to stimuli with a positive or negative valence (unconditioned stimulus, US). The total duration of the CE is approximately 15 minutes.

SUMMARY:
The hypothesis is that, compared to those in the control group (i.e., diet-related evaluative conditioning), participants in the Physical Activity (PA) group (i.e. PA-friendly evaluative conditioning) will exhibit (1) a higher intensity (power setting) on an ergocycle during a free Physical Activity session in their rehabilitation program and (2) A greater increase in the implicit attitude score.

The primary objective will be to evaluate the effect of evaluative conditioning (EC) on the intensity of physical activity produced by post-myocardial infarction patients involved in a cardiac rehabilitation program.The secondary objective of this study will be to evaluate the mediating effect of implicit attitude change in the effect of evaluative conditioning on adopted behaviors.

DETAILED DESCRIPTION:
More specifically, post-myocardial infarction physical activity has been shown to reduce cardiac morbidity and mortality. Indeed, exercise improves cardiovascular health through mechanisms such as lowering blood pressure, weight reduction, and increased insulin sensitivity. Although there are no formal guidelines for physical activity (PA) after Myocardial Infarction, patients are encouraged to achieve 150 minutes of low-to-moderate intensity PA per week.

Nevertheless, despite the growing body of scientific evidence and the widespread dissemination of information about the benefits of PA, the recommendations have been difficult for post-myocardial infarction patients to comply with. There is evidence to suggest that post-cardiac rehabilitation patients struggle to maintain sustained PA. This may be due to a number of barriers, including fatigue, mood disorders, a lack of motivation, or kinesiophobia.

Continued improvements in monitoring physical activity and the development of policies and programs to increase activity levels appears to be a necessity. This may reduce the burden of physical inactivity and noncommunicable diseases (eg, cardiovascular disease). Therefore, one of the major challenges is to succeed in identifying the main determinants playing a role in the lack of adoption of regular PA. Indeed, targeting these determinants would ultimately allow us to improve the PA promotion strategies already in place for the population. However, maintenance of a practice over time is a complex issue that may be influenced by a multitude of factors. Among these, previous work suggests that the identification of motivational determinants of physical activity represents a relevant research object in this context.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have given written informed consent to participate in the trial
* Patients must be aged18 to 75 years old
* It must be less than 6 months after a first episode of myocardial infarction treated medically or by revascularization

Exclusion Criteria:

* Patients with a disability preventing the performance of a bimanual test or an ergocycle task
* Patients who are unable to give written informed consent or who have refused to sign the consent form

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Post-myocardial infarction patients involved in a cardiac rehabilitation program at Nîmes University Hospital, France.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Effect of evaluative conditioning on the intensity of physical activity produced by post-myocardial infarction patients involved in a cardiac rehabilitation program. Control group | Day 0 before completing the Implicit Association Test
  The choice of intensity (power setting) on the ergocycle will be measured by controlling it before the Evaluative Conditioning procedure.the ergocycle task consists of pedaling on an indoor bicycle for about 15 minutes, we will only be interested in the intensity data of this task (This task is an integral part of the patients' care at the University Hospital and will be supervised by health professionals - physiotherapist, physical activity teachers, etc.)
Effect of evaluative conditioning on the intensity of physical activity produced by post-myocardial infarction patients involved in a cardiac rehabilitation program. Control group | Day 0 after completing the Implicit Association Test
  The choice of intensity (power setting) on the ergocycle will be measured by controlling it before the Evaluative Conditioning procedure.the ergocycle task consists of pedaling on an indoor bicycle for about 15 minutes, we will only be interested in the intensity data of this task (This task is an integral part of the patients' care at the University Hospital and will be supervised by health professionals - physiotherapist, physical activity teachers, etc.)
Effect of evaluative conditioning on the intensity of physical activity produced by post-myocardial infarction patients involved in a cardiac rehabilitation program. Experimental group | Day 0 before completing the Implicit Association Test
  The choice of intensity (power setting) on the ergocycle will be measured by controlling it before the Evaluative Conditioning procedure.the ergocycle task consists of pedaling on an indoor bicycle for about 15 minutes, we will only be interested in the intensity data of this task (This task is an integral part of the patients' care at the University Hospital and will be supervised by health professionals - physiotherapist, physical activity teachers, etc.)
Effect of evaluative conditioning on the intensity of physical activity produced by post-myocardial infarction patients involved in a cardiac rehabilitation program. Experimental group | Day 0 after completing the Implicit Association Test
  The choice of intensity (power setting) on the ergocycle will be measured by controlling it before the Evaluative Conditioning procedure. Note that the ergocycle task consists of pedaling on an indoor bicycle for about 15 minutes, (this task is an integral part of the patients' care at the University Hospital and will be supervised by health professionals - physiotherapist, physical activity teachers, etc.). Only the intensity data of this task will be recorded

SECONDARY OUTCOMES:
Mediating effect of implicit attitudinal change in the effect of evaluative conditioning on adopted behaviors. Control group | Time 0, before taking the test
  The change in implicit attitudes will be measured by comparing the Implicit Association Test pretest score (T0) and the Implicit Association Test posttest score (T1).
Mediating effect of implicit attitudinal change in the effect of evaluative conditioning on adopted behaviors. Experimental group | Time 0, before taking the test
  The change in implicit attitudes will be measured by comparing the Implicit Association Test pretest score (T0) and the Implicit Association Test posttest score (T1)
Mediating effect of implicit attitudinal change in the effect of evaluative conditioning on adopted behaviors. Control group | Time 0, after taking the test
  The change in implicit attitudes will be measured by comparing the Implicit Association Test pretest score (T0) and the Implicit Association Test posttest score (T1)
Mediating effect of implicit attitudinal change in the effect of evaluative conditioning on adopted behaviors. Experimental group | Time 0, after taking the test
  The change in implicit attitudes will be measured by comparing the Implicit Association Test pretest score (T0) and the Implicit Association Test posttest score (T1)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamer M, O'Donovan G, Murphy M. Physical Inactivity and the Economic and Health Burdens Due to Cardiovascular Disease: Exercise as Medicine. Adv Exp Med Biol. 2017;999:3-18. doi: 10.1007/978-981-10-4307-9_1. PMID 29022254
- [Background] Clark AM, Hartling L, Vandermeer B, McAlister FA. Meta-analysis: secondary prevention programs for patients with coronary artery disease. Ann Intern Med. 2005 Nov 1;143(9):659-72. doi: 10.7326/0003-4819-143-9-200511010-00010. PMID 16263889
- [Background] Birtwistle SB, Jones I, Murphy R, Gee I, Watson PM. "Do what you can with a happy heart": a longitudinal study of patient and family members' lived experiences of physical activity post-myocardial infarction. Disabil Rehabil. 2022 Jul;44(14):3661-3670. doi: 10.1080/09638288.2021.1878560. Epub 2021 Mar 1. PMID 33646893
- [Background] Karmali KN, Davies P, Taylor F, Beswick A, Martin N, Ebrahim S. Promoting patient uptake and adherence in cardiac rehabilitation. Cochrane Database Syst Rev. 2014 Jun 25;(6):CD007131. doi: 10.1002/14651858.CD007131.pub3. PMID 24963623
- [Background] Antoniewicz F, Brand R. Learning to Like Exercising: Evaluative Conditioning Changes Automatic Evaluations of Exercising and Influences Subsequent Exercising Behavior. J Sport Exerc Psychol. 2016 Apr;38(2):138-48. doi: 10.1123/jsep.2015-0125. Epub 2016 Mar 15. PMID 27385674
- [Background] Chevance G, Bernard P, Chamberland PE, Rebar A. The association between implicit attitudes toward physical activity and physical activity behaviour: a systematic review and correlational meta-analysis. Health Psychol Rev. 2019 Sep;13(3):248-276. doi: 10.1080/17437199.2019.1618726. Epub 2019 Jun 12. PMID 31117901
- [Background] Rebar AL, Dimmock JA, Jackson B, Rhodes RE, Kates A, Starling J, Vandelanotte C. A systematic review of the effects of non-conscious regulatory processes in physical activity. Health Psychol Rev. 2016 Dec;10(4):395-407. doi: 10.1080/17437199.2016.1183505. Epub 2016 May 20. PMID 27118430
- [Background] Hofmann W, De Houwer J, Perugini M, Baeyens F, Crombez G. Evaluative conditioning in humans: a meta-analysis. Psychol Bull. 2010 May;136(3):390-421. doi: 10.1037/a0018916. PMID 20438144
- [Background] Rogerson MC, Murphy BM, Bird S, Morris T. "I don't have the heart": a qualitative study of barriers to and facilitators of physical activity for people with coronary heart disease and depressive symptoms. Int J Behav Nutr Phys Act. 2012 Nov 30;9:140. doi: 10.1186/1479-5868-9-140. PMID 23194091
- [Background] Rhodes RE, Janssen I, Bredin SSD, Warburton DER, Bauman A. Physical activity: Health impact, prevalence, correlates and interventions. Psychol Health. 2017 Aug;32(8):942-975. doi: 10.1080/08870446.2017.1325486. Epub 2017 May 30. PMID 28554222